CLINICAL TRIAL: NCT02520219
Title: The Efficacy and Safety Research of Endostar Combined With GDP to Treat Aggressive Peripheral T-cell Lymphoma (PTCL) in Phase II Clinical Study.
Brief Title: Endostar Aggressive Treatment of Peripheral T-cell Lymphoma (PTCL) Phase II Clinical Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing NingQi Medicine Science and Technology Co., Ltd. (Industry)
Collaborators: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Endostar-PTLC-001
Record Dates: First submitted 2015-07-26; First posted 2015-08-11 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Peripheral T-cell Lymphomas
Keywords: Peripheral T-cell lymphomas,Endostar
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Guanosine Diphosphate; endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GDP+Endostar (Experimental): Patients in this group will be given conventional chemotherapy medicine:
  GDP (gemcitabine+dexamethasone+cis-platinum)chemotherapy by treatment guidelines for Peripheral T-cell Lymphoma and Endostar.
  Interventions: Drug: GDP; Biological: Endostar
- GDP (Active Comparator): Patients in this group will be given conventional chemotherapy medicine:
  GDP (gemcitabine+dexamethasone+cis-platinum) chemotherapy by treatment guidelines for Peripheral T-cell Lymphoma.
  Interventions: Drug: GDP

INTERVENTIONS:
Drug: GDP — GDP is a a combination therapy,repeated every 21 days. GEM(gemcitabine)1000mg/m2,ivgtt,30,d1、8; DXM(dexamethasone),40mg/d,p.o,d1-4; DDP(cis-platinum),75mg/m2,ivgtt,>1h,d1; or DDP25 mg/m2,ivgtt,>1h,d1-3.
Biological: Endostar — Endostar is a continuous intravenous injection pump, continuous intravenous pumped by seven consecutive days,d1- d7, which is 168 hours .Endostar pumping well dose is 30 mg every 24 hours.
  Repeated every 21 days.
  Arms: GDP+Endostar

SUMMARY:
The aim of this study is to evaluate anti-tumor safety and efficacy of endostar®（Human recombinant endostatin injection）combined with traditional GDP （gemcitabine+dexamethasone+cis-platinum）chemotherapy for newly diagnosed or relapsed PTCL(aggressive peripheral T-cell lymphomas) patients in phase II clinical study.

DETAILED DESCRIPTION:
Endostar is a conventional drug for treatment of advanced non-small cell lung cancer, nowadays,Endostar has been used in a variety of extra-pulmonary tumor treatment in clinical.Some basic experiments and clinical researchs confirm that Endostar can restitute the tumor stability after cyclophosphamide or rituximab treatment.

The aim of this study is to evaluate anti-tumor safety and efficacy of endostar for newly diagnosed or relapsed PTCL patients based on chemotherapy combined with conventional GDP.This is a multi-center, open, randomized-controlled, phase II clinical study.

Following a run-in period, approximately 60 subjects will be randomly assigned to conventional chemotherapy treatment group, endostar and conventional chemotherapy treatment group for 1 year. After the 1 year treatment period, subjects in two treatments arms will be followed for 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed or relapsed PTCL patients by pathology, and / or cytology examination, which are required to receive chemotherapy;
2. At least 1 single size measurable lesions, CT, MRI, Bultrasound scan or PET-CT scan shows more than 15mm；
3. Physical condition is good: ECOG score between 0-2 points；
4. The expected survival time is more than 3 months；
5. Age 18 years or older,unlimited gender；
6. Fit chemotherapy indications and basic requirements, including normal peripheral hemogram,no obvious abnormal function of heart, liver and kidney, normal ECG;no great trauma without healing；

   The test indicators must fit the following requirements:

   Cardiac ultrasound LVEF≥50%； Peripheral blood：WBC≥3.5×109/L，PLT≥70×109/L，Hb≥80g/L Renal function：Cr≤2.0×UNL（Upper limit of normal value） Liver function：BIL≤2.0×UNL，ALT/AST≤2.5×UNL
7. No serious allergic reaction to biological agents, especially E. coli gene engineering products；
8. Voluntary participation, good compliance, cooperate with the experimental observation, and sign a written informed consent。

Exclusion Criteria:

1. Inert T cell lymphoma (such as mycosis fungoides /Sezary syndrome), ALK positive anaplastic large cell lymphoma；
2. Patients who received chemotherapy drugs in the past;
3. Pregnant women,lactating women,or having fertility but not taking contraceptive measures；
4. Patients with serious uncontroled acute infection;or suppurative and chronic infection and unhealing wound；
5. Patients with original serious heart disease, including: high-risk cardiac arrhythmias of congestive heart failure,uncontroled instability angina, myocardial infarction and severe heart valve disease and intractable hypertension；
6. Patients with less control of the nervous, mental illness or mental disorders, poor compliance, and the description of the treatment response；
7. Patients with primary central nervous system lymphoma or lymphoma involving central nervous system；
8. Patients with abnormal coagulation function and severe thrombosis;
9. Patients who participated in other clinical trials；
10. The researchers considered that patients should not be in this trial。

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
ORR(Overall release rate) | Change from Baseline at the week 6,12, 18 of treatment phase and the month 3, 6, 9 and 12, 15, 18, 21, 24, 27, 30 ,33,36 of the followup phase
  According to the Cheson standard recommended by NCCN (National Comprehensive Cancer Network)guidelines of USA, the evaluation of the clinical effect of the drug on tumor was evaluated by comparing the change of tumor size and duration.

SECONDARY OUTCOMES:
PFS（progression-free survival） | Change from Baseline at the week 3, 6, 9, 12, 15,18 of the treatment phase, the month 3, 6, 9 and 12, 15, 18, 21, 24, 27, 30 ,33,36 of the followup phase.
DCR(disease control rate) | Change from Baseline at the week 3, 6, 9, 12, 15,18 of the treatment phase, the month 3, 6, 9 and 12, 15, 18, 21, 24, 27, 30 ,33,36 of the followup phase.
OS（overall survival） | Change from Baseline at the week 3, 6, 9, 12, 15,18 of the treatment phase, the month 3, 6, 9 and 12, 15, 18, 21, 24, 27, 30 ,33,36 of the followup phase.
Adverse reaction | Change from Baseline at the week 3, 6, 9, 12, 15,18 of the treatment phase
The quality of life（QOL） Questionnaire | Change from Baseline at the week 3, 6, 9, 12, 15,18 of the treatment phase, the month 3, 6, 9 and 12, 15, 18, 21, 24, 27, 30 ,33,36 of the followup phase.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu province tumor hospital, Nanjing, Jiangsu, China